CLINICAL TRIAL: NCT03840577
Title: Effect of Bispectral Index (BIS)-Guided Sedation on Delirium and Sedative Drug Requirements in Critically Ill Patients Under Deep Sedation
Brief Title: BIS-Guided Sedation in Critically Ill Patients Under Deep Sedation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Ivan A Huespe, MD, Principal Investigator, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3880
Record Dates: First submitted 2019-02-03; First posted 2019-02-15 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Delirium; Sedative Overdose
Keywords: Deep Sedation; Bispectral index; Critical care patients; Delirium; Sedatives
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: Patients will be assigned according to the randomization to clinical monitoring groups or Bispectral Index (BIS) monitoring group. The ranzomization will be stratified randomization by neuromuscular bloquers.
Who Masked: Participant, Outcomes Assessor
Masking Description: The primary outcome "Compare delirium and coma-free days until 14 days after the end of deep sedation" will be assessed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) scale. The evaluations will be conducted by blinded evaluators who are unaware of the patient's assigned sedation management group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sedation guided by Clinical Scales (No Intervention): Sedative guided by RASS (Richmond Agitation-Sedation Scale) score. Target RASS: -4 / -5.
- Sedation guided by Bispectral Index (Experimental): Sedation guided by the Bispectral Index (BIS). Target BIS between 40 to 60.
  Interventions: Device: Monitorization of sedation by Bispectral Index

INTERVENTIONS:
Device: Monitorization of sedation by Bispectral Index — The sedative dose administered through a continuous infusion pump will be adjusted based on the BIS value to maintain a target range of 40 to 60. If the BIS value is below the target range, the dose will be increased, and if it exceeds the range, the dose will be decreased, aiming to keep the BIS within the desired range.
  Arms: Sedation guided by Bispectral Index

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of sedation guided by the bispectral index (BIS) in reducing the incidence of delirium and the doses of sedative drugs used in critical patients who require deep sedation. The main questions this study aims to answer are:

* Does sedation guided by BIS lead to higher delirium and coma-free days compared to clinical monitoring?
* Does sedation guided by BIS result in reduced doses of sedative drugs compared to clinical monitoring?

Participants in this study will be randomly assigned to one of two groups:

Clinical Monitoring Group: Participants in this group will receive sedation based on clinical scales. These participants will also be fitted with a BIS sensor, but the sensor will be covered.

Sedation Guided by BIS Group: Participants in this group will receive sedation guided by the bispectral index.

The study will be conducted as a prospective, controlled, blind intervention trial with random distribution and intention to treat. The primary outcomes to be evaluated include:

* Delirium and coma-free days after the end of deep sedation using the Confusion Assessment Method for the ICU (CAM-ICU) scale.
* Total dose of sedative drugs administered.
* BIS values

Researchers will compare the two groups to determine if sedation guided by BIS is associated with a higher number of delirium and coma-free days, reduced sedative drug doses, and higher values of BIS compared to clinical monitoring.

DETAILED DESCRIPTION:
A Phase 4, randomized (1:1), controlled, double-blind, unicenter clinical trial aims to assess the effectiveness of sedation guided by the Bispectral Index (BIS) compared to sedation guided by clinical scales in critically ill patients under deep sedation. The primary objective is to investigate whether BIS-guided sedation can reduce the incidence of delirium and decrease the doses of sedative drugs administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Under mechanical ventilation in the intensive care unit
* Indication of deep sedation (RASS objective -4, -5)
* Admission to the ICU or indication of deep sedation up to 8 hours prior to randomization.

Exclusion Criteria:

* Patients with end-of-life care.
* Family refusal to participate in the study.
* Impossibility to place the BIS sensor (burns, extensive lesions on the forehead, prone position, etc.).
* Patients with intracranial hypertension or convulsive status, in whom sedation has the objective of suppressing electroencephalographic waves.
* Patients who, following a decrease in sedation, have a coma, vegetative state or a state of minimal consciousness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Compare delirium and coma free days until 14 days after end of deep sedation | Up to 14 days post end of deep sedation
  To compare the number of Delirium and Coma-Free Days until day 14 after the cessation of deep sedation in patients receiving sedation guided by the Bispectral Index (BIS) vs. sedation guided by clinical scales. Delirium will be assessed using the CAM-ICU scale (Ely EW et al.) by non-ICU researchers who are blinded to the randomization allocation. The delirium evaluation will begin when the patient reaches a Richmond Agitation-Sedation Scale (RASS) score of > -3.
Compare the doses of sedative drugs received | From date of randomization until the date of end of deep sedation or date of death from any cause, whichever came first, assessed up to 90 days
  To compare the total doses of Propofol, Midazolam, and Remifentanil (calculated in mg/kg) received during the period of deep sedation
Compare values of BIS | From date of randomization until the date of end of deep sedation or date of death from any cause, whichever came first, assessed up to 90 days
  To compare the values of Bispectral Index (BIS) in patients receiving sedation guided by the Bispectral Index (BIS) versus sedation guided by clinical scales. This outcome will assess the BIS values recorded during the period of deep sedation and compare them between the two groups

SECONDARY OUTCOMES:
Time with values of BIS less than 40 | From date of randomization until the date of end of deep sedation or date of death from any cause, whichever came first, assessed up to 90 days
  To compare the number of hours that patients receiving sedation guided by the Bispectral Index (BIS) vs. sedation guided by clinical scales had registered Bispectral Index (BIS) values below 40 during the period of deep sedation. The duration of time with BIS values below 40 will be recorded for each patient.
Compare days alive and free of the ICU | From date of randomization until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 120 days
  To compare the effect of sedation guided by the Bispectral Index (BIS) vs. sedation guided by clinical scales on days alive and free of the ICU
Compare days alive and free of the hospital | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 120 days
  To compare the effect of sedation guided by the Bispectral Index (BIS) vs. sedation guided by clinical scales on days alive and free of the hospital
Compare days alive and free of mechanical ventilation through Study Day 30 | From date of randomization until the date of end of mechanical ventilation or date of death from any cause, whichever came first, assessed up to 30 days
  To compare the effect of sedation guided by the Bispectral Index (BIS) vs. sedation guided by clinical scales on the number of days alive and free of mechanical ventilation through Study Day 30
Compare days alive and free of mechanical ventilation through Study Day 60 | From date of randomization until the date of end of mechanical ventilation or date of death from any cause, whichever came first, assessed up to 60 days
  To compare the effect of sedation guided by the Bispectral Index (BIS) vs. sedation guided by clinical scales on the number of days alive and free of mechanical ventilation through Study Day 60
Compare delirium and coma free days until 14 days after end of deep sedation in patients who had more than 24 hours of deep sedation | Up to 14 days post end of deep sedation
  To compare the number of Delirium and Coma-Free Days until day 14 after the cessation of deep sedation in patients receiving sedation guided by the Bispectral Index (BIS) vs. sedation guided by clinical scales. Delirium will be assessed using the CAM-ICU scale (Ely EW et al.) by non-ICU researchers who are blinded to the randomization allocation. The delirium evaluation will begin when the patient reaches a Richmond Agitation-Sedation Scale (RASS) score of > -3, in patients who had more than 24 hours of deep sedation

OTHER OUTCOMES:
Compare mortality at 60 days after randomization | Until 60 days after randomization
  To compare the effect of sedation guided by the Bispectral Index (BIS) vs. sedation guided by clinical scales on mortality at 60 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giannasi, MD, Study Chair — Hospital Italiano de Buenos Aires; Federico Carini, MD, Study Director — Hospital Italiano de Buenos Aires; Ivan A. Huespe, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Capital Federal, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available upon reasonable request.
Supporting Information: Analytic Code
Time Frame: The data will be made available at the end of the study, in 2024.
Access Criteria: All data requirements will be evaluated by the principal investigator and the local Institutional Review Board to ensure compliance with ethical and regulatory guidelines regarding data access and protection

REFERENCES:
- [Background] MacKenzie KK, Britt-Spells AM, Sands LP, Leung JM. Processed Electroencephalogram Monitoring and Postoperative Delirium: A Systematic Review and Meta-analysis. Anesthesiology. 2018 Sep;129(3):417-427. doi: 10.1097/ALN.0000000000002323. PMID 29912008
- [Background] Salluh JI, Soares M, Teles JM, Ceraso D, Raimondi N, Nava VS, Blasquez P, Ugarte S, Ibanez-Guzman C, Centeno JV, Laca M, Grecco G, Jimenez E, Arias-Rivera S, Duenas C, Rocha MG; Delirium Epidemiology in Critical Care Study Group. Delirium epidemiology in critical care (DECCA): an international study. Crit Care. 2010;14(6):R210. doi: 10.1186/cc9333. Epub 2010 Nov 23. PMID 21092264
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Shetty RM, Bellini A, Wijayatilake DS, Hamilton MA, Jain R, Karanth S, Namachivayam A. BIS monitoring versus clinical assessment for sedation in mechanically ventilated adults in the intensive care unit and its impact on clinical outcomes and resource utilization. Cochrane Database Syst Rev. 2018 Feb 21;2(2):CD011240. doi: 10.1002/14651858.CD011240.pub2. PMID 29464690
- [Derived] Huespe I, Giunta D, Acosta K, Avila D, Prado E, Sanghavi D, Bisso IC, Giannasi S, Carini FC. Comparing Bispectral Index Monitoring vs Clinical Assessment for Deep Sedation in the ICU: Effects on Delirium Reduction and Sedative Drug Doses-A Randomized Trial. Chest. 2024 Oct;166(4):733-742. doi: 10.1016/j.chest.2024.05.031. Epub 2024 Jun 18. PMID 38901489